CLINICAL TRIAL: NCT00773916
Title: The Role of Adverse Environment Factors, Family Functioning and Parental Psychopathology in the Response to Treatment With Methylphenidate in Children and Adolescents With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Luis Augusto Rohde MD, Federal University of Rio Grande do Sul
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06-208
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder; Attention Deficit Disorders with Hyperactivity; Hyperkinetic Syndrome; Family Function; Adverse Factors; Parental Psychopathology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methylphenidate — Dose increments according to clinical evaluation, starting with 0,3 mg/kg of weight/day

SUMMARY:
The purpose of this study is to investigate the association of adverse environmental factors, parental psychopathology, family functioning and genetic factors and the response to methylphenidate treatment in children and adolescents with Attention Deficit/Hyperactivity Disorder.

DETAILED DESCRIPTION:
Attention Deficit/Hyperactivity Disorder (ADHD) is a chronic disorder, with a worldwide estimated prevalence of 5,29%. It is associated with a high risk of functional impairment in many aspects of the patient´s life, such as academic achievements, peers relationships and physical injuries. There are few studies assessing predictive factors of clinical response to treatment. Different patterns of family functioning, such as high family conflict and low family cohesion might be associated with a poor treatment response, possibly mediating the effects of higher severity af the disorder and/or higher prevalence of comorbidity. Parental psychopathology has been associated with a poorer prognosis and is related with family functioning. Adverse social factors have long been studied and are associated with an increased risk for general mental disease, including ADHD, as well as a poorer prognosis. Different genetic factors have been studied and associated with different aspects of the disorder and different clinical responses to treatments. There are no studies evaluating how those factors interact with each other in a Brazilian population.

ELIGIBILITY:
Inclusion Criteria:

* ADHD
* Age: 5 - 18
* Primary Indication of Methylphenidate

Exclusion Criteria:

* IQ < 70
* Clinical conditions that preclude use of methylphenidate

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
SNAP -IV scores | 1, 2, 3 and 6 months of treatment
CGI scores | 1, 2, 3 and 6 months of treatment

SECONDARY OUTCOMES:
Scores in CGAS | 1, 2, 3 and 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Rohde, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- ADHD Outpatient Program - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- See also: Related Info — http://www6.ufrgs.br/prodah/